CLINICAL TRIAL: NCT05709431
Title: A Prospective, Monocentric, Open, Non-controlled Study Evaluating the French Version of the CIQoL-35 Quality of Life Questionnaire in Adult Cochlear Implant Use
Brief Title: A Study Evaluating the French Version of the CIQoL-35 Quality of Life Questionnaire in Adult Cochlear Implant Use.
Acronym: CIQoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: OM26
Record Dates: First submitted 2022-10-12; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: PROM; Cochlear Hearing Loss; Hearing Loss; Quality of Life
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire CIQoL-35 — The Cochlear Implant - Quality of Life (CIQoL) PROM is a quality-of-life assessment questionnaire for adults with cochlear implants (1-7). The CIQoL responds to an important need for a questionnaire that captures the benefits of cochlear implantation as perceived by patients and that can be used in clinical practice. The CIQoL is available in two lengths: 35 questions (CIQoL-35) and 10 questions (CIQoL-10). The CIQoL-35 has interesting measurement properties including good construct validity, convergent validity, and test-retest reliability.

SUMMARY:
The Cochlear Implant - Quality of Life (CIQoL) PROM is a quality-of-life assessment questionnaire for adults with cochlear implants. The CIQoL responds to an important need for a questionnaire that captures the benefits of cochlear implantation as perceived by patients and that can be used in clinical practice.

DETAILED DESCRIPTION:
The CIQoL-35 has been translated and adapted from English to French in accordance with the guidelines of Hall and colleagues.

The purpose of the current study is to describe the measurement properties of the French CIQoL-35 questionnaire.

Hall et al recommend that at least 8 patients participate in any qualitative testing of the translation (n=13 in the previous study) and that at least 50 patients participate in a measurement property evaluation (n=50 in the present study).

The aim of this study is not to assess the performance of the device or compare the performance of different devices/brands but to correlate quality of life scores with speech understanding in patients with cochlear implants. The main objective of the study is to validate the translation of the questionnaire, the correlation is a secondary criterion.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) user of at least one cochlear implant system,
* Duration of cochlear experience ≥ 6 months (period from cochlear implant activation to study enrolment),
* Psychological/literacy ability to read, understand, and complete the questionnaire.

Exclusion Criteria:

* Patient who participated in initial validation of the French CIQoL-35 (CIQoL project part 1),
* Patient with a psychological or linguistic inability to understand the information sheet or the questionnaire,
* Patient under legal protection or deprived of liberty,
* Unwillingness or inability to comply with all investigational requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients aged 18 years and older, with bilateral, severe-to-profound sensorineural hearing loss, with at least one cochlear implant for more than 6 months with the ability to read, understand, and indicate their answers to the 35-item French CIQoL questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the measurement properties of the French CIQoL-35. | Day 1 (one visit planned)
  The patient is given a paper questionnaire containing the 35 items. The questionnaire indicates the following instructions:
  "Think about your daily life with your cochlear implant (and/or hearing aid, if you also use one). Answer how often each of the following statements applies to your feelings and experiences. Answer how often each statement applies even if you don't use cochlear implants or hearing aids."

SECONDARY OUTCOMES:
Speech performance in quiet | Day 1 (one visit planned)
  Speech perception performance in sound field in best-aided condition (i.e., using a contralateral hearing aid if the patient does on a daily basis): Score at Lafon test (in words/phonemes) on 2 lists: 8 and 19 at 60 dB A in quiet (15 min)
Speech performance in noise | Day 1 (one visit planned)
  Score at VRB test
Describe the duration of French CIQoL-35 administration | Day 1 (one visit planned)
  Measure of duration (in minutes) to complete the CIQoL-35 done by the audiologist with a timer. The CIQoL questionnaire present 35 questions with 6 subscales with established validity; the CIQOL-35 takes 4.5 minutes to complete. For each question, the patient have 5 response options (Never (lowest score), Rarely, Sometimes, Often, Always (higher score)).
Correlation between variable of interest CIQoL score and explicative variable such as speech performance and demographics. | Day 1 (one visit planned)
  Correlation between variable of interest CIQoL score and explicative variable such as speech performance and demographics

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MOSNIER, Principal Investigator — GH Pitié-Salpêtrière, APHP Sorbonne Université, Paris, France
Locations (1):
- Centre de Recherche en Audiologie adulte, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided